CLINICAL TRIAL: NCT00253084
Title: A Randomized, Double-Blind, Cross-Over Study to Compare IPX054 to Carbidopa-Levodopa Immediate-Release Tablets in Subjects With Parkinson's Disease
Brief Title: Comparison of IPX054 and Immediate-Release Carbidopa-Levodopa in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IPX054-B04-07
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2017-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPX054 - CD-LD IR (Other): Subjects received IPX054 200 mg b.i.d and CD-LD IR Placebo q.i.d for 2 weeks and then received IPX054 Placebo b.i.d and CD-LD IR q.i.d for 2 weeks.
  Interventions: Drug: IPX054 200 mg; Drug: CD-LD IR; Drug: IPX054 Placebo; Drug: CD-LD IR Placebo
- CD-LD IR - IPX054 (Other): Subjects received IPX054 Placebo b.i.d and CD-LD IR q.i.d for 2 weeks and then IPX054 200 mg b.i.d and CD-LD IR Placebo q.i.d for 2 weeks.
  Interventions: Drug: IPX054 200 mg; Drug: CD-LD IR; Drug: IPX054 Placebo; Drug: CD-LD IR Placebo

INTERVENTIONS:
Drug: IPX054 200 mg — IPX054 containing 50 mg carbidopa and 200 mg levodopa
  Other Names: CD-LD ER 200 mg
Drug: CD-LD IR — CD-LD IR containing 25 mg carbidopa and 100 mg levodopa
Drug: IPX054 Placebo — Placebo to match IPX054 200 mg
Drug: CD-LD IR Placebo — Placebo to match CD-LD IR

SUMMARY:
The purpose of this study is to compare the clinical efficacy of IPX054 to immediate-release carbidopa-levodopa in subjects with Parkinson's disease.

DETAILED DESCRIPTION:
IPX054 contains two different drugs called levodopa and carbidopa in one tablet.

* levodopa turns into a material called 'dopamine' in your brain. The dopamine helps to improve the symptoms of your Parkinson's disease.
* carbidopa belongs to a group of medicines called 'aromatic amino acid decarboxylase inhibitors'. It helps levodopa work more effectively by slowing the speed at which levodopa is broken down in your body.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's disease based on CAPIT (Core Assessment Program for Intracerebral Transplantations) criteria.
* Currently being treated with immediate-release carbidopa-levodopa with a stable dosing regimen over the past 4 weeks.

Exclusion Criteria:

* Diagnosed with atypical parkinsonism.
* Allergic or non-responsive to previous carbidopa-levodopa therapy.
* Active or history of narrow-angle or wide-angle glaucoma.
* History of seizure or epilepsy, or is currently taking an anti-convulsant for treatment of seizure.
* Requires concomitant therapy with tricyclic antidepressants, MAO-B inhibitors, COMT inhibitors or anticholinergics.
* Treatment with any neuroleptic agent, including atypical neuroleptics, within the previous 6 months.
* Treatment with any dopaminergic blocking agent within the previous 6 months.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
"ON" time without disabling dyskinesias | 2 weeks

SECONDARY OUTCOMES:
UPDRS analysis | 2 weeks
Mean time to "ON" | 2 weeks
Mean time to "wearing OFF" | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (2):
- United States (2):
  - Site 1, Chicago, Illinois
  - Site 2, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No